CLINICAL TRIAL: NCT00132951
Title: A Randomized, Investigator Blinded, Multi-Center Clinical Study To Compare Patient Outcomes and Clinical Effectiveness of Telithromycin Versus Azithromycin in Outpatients With Lower Respiratory Tract Infections
Brief Title: KEYS: Study Comparing Clinical Health Outcomes of Telithromycin Versus Azithromycin in Outpatients With Community-acquired Lower Respiratory Tract Infections
Acronym: KEYS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMR3647A_4019
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2009-08

CONDITIONS: Respiratory Tract Infections; Chronic Bronchitis; Pneumonia
MeSH Terms: conditions — Respiratory Tract Infections; Bronchitis, Chronic; Pneumonia | interventions — telithromycin; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Telithromycin — Telithromycin (AECB: 2 tablets per day for Days 1-5; CAP: 2 tablets per day for Days 1-7)
  Other Names: Ketek
Drug: Azithromycin — Azithromycin (AECB: 2 tablets on Day 1 then 1 tablet + 1 placebo tablet per day for Days 2-5; CAP: 2 tablets on Day 1 then 1 tablet + 1 placebo tablet per day for Days 2-5 then 2 placebo tablets per day for Days 6-7)

SUMMARY:
The purpose of this study is to determine if 1 course of antibiotic treatment with telithromycin is superior to azithromycin in the treatment of lower respiratory tract infections (LRTIs), acute exacerbations of chronic bronchitis (AECBs) and community-acquired pneumonia (CAP) in the community setting.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria will be considered for enrollment into the study:

* Male and female adult outpatient subjects diagnosed with AECB or CAP
* Female subjects must be either postmenopausal for ≥ 1 year or surgically incapable of bearing children. Women of childbearing potential must have a normal menstrual flow ≤ 1 month before study entry, a negative serum pregnancy test immediately prior to study entry, and meet the criteria for acceptable birth control.
* Informed consent must be obtained in writing for all subjects upon enrollment.
* Subjects will have a diagnosis of AECB or CAP, as defined below.

AECB-Specific Inclusion Criteria:

* Subjects greater than or equal to 35 years of age
* Subjects with a documented history of chronic bronchitis: with a basal forced expiratory volume in one second (FEV1) < 70% and > 35%; who have had at least one or more AECB in the previous year; and with FEV1/forced vital capacity (FVC) < 70%.
* Subjects with a clinical diagnosis of AECB, presumed to be due to bacterial infection based on increased sputum purulence with either increased dyspnea or sputum volume
* Subjects producing spontaneous sputum
* Subjects with a ≥ 10 pack-year history of cigarette smoking

CAP-Specific Inclusion Criteria:

* Fever (oral temperature > 38°C [100.4°F] or tympanic temperature > 38.5°C [101.2°F] or rectal temperature > 39°C [102.2°F])
* Chills
* Pleuritic chest pain
* Cough
* Spontaneous production of purulent sputum or a change in sputum character
* Auscultatory findings (such as rales [also known as crepitations] and/or evidence of pulmonary consolidation [ie, dullness on percussion, bronchial breath sounds, egophony])
* Subjects greater than or equal to 18 years of age
* Chest x-ray findings that support a clinical diagnosis of bacterial pneumonia (eg, presence of presumably new infiltrate[s])
* Subjects with a clinical diagnosis of mild to moderate CAP due to bacterial infection based on at least 1 of the following signs and symptoms of CAP:
* In addition, subjects with a clinical diagnosis of CAP will have at least 1 of the following signs and symptoms of CAP:

  * Dyspnea or tachypnea (particularly if progressive in nature)

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

* Subjects with a known history of congenital long-QTc syndrome
* Subjects who are pregnant or breast-feeding
* Subjects who have hypersensitivity to telithromycin, azithromycin, or the macrolide classes of antibiotics
* Subjects who require or receive treatment with rifampin (Rifadin), phenytoin (Dilantin), carbamazepine (Carbatrol, Tegretol), phenobarbital, or St. John's wort (herbal supplement) within 2 weeks prior to Visit 1 or during the study
* Subjects who require treatment during the study with ergot alkaloid derivatives, cisapride (Propulsid), pimozide (Orap), bromocriptine, cabergoline (Dostinex), or pergolide (Permax)
* Subjects who have previously participated in this study
* Subjects with a previous history of myasthenia gravis
* Subjects with current acute respiratory failure or subjects who require aggressive airway management
* Hospitalized subjects and subjects from institutional care facilities
* Subjects who have been treated with oral or parenteral antibiotics within 14 days prior to enrollment or who plan to take antibiotics other than study drug during the treatment period
* Subjects who are receiving other medications, including systemic antimicrobial agents, or who have other disease conditions or infections that could interfere with the evaluation of drug efficacy or safety
* Subjects with a concomitant condition (including clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease) that makes either implementation of the protocol or interpretation of the study results difficult
* Subjects with a progressively fatal disease or life expectancy of < 3 months
* Subjects who have received any other investigational drug or device within 1 month prior to study entry, or who have such treatment planned during the study period
* Subjects with a recent (within 3 months) history of drug or alcohol abuse
* Immunocompromised subjects, including but not limited to subjects with: known human immunodeficiency virus infection (CD4 count < 200/mm3); known neutropenia (< 1500 neutrophils/mm3); chronic corticosteroid therapy (≥ 10 mg/day prednisolone therapy or equivalent for at least the past 3 months); immunosuppressant treatment, other than corticosteroids, within the previous 6 months; splenectomized subjects or subjects with known hyposplenia or asplenia.
* Subjects with mental conditions that render them unable to understand the nature, scope, and possible consequences of the study
* Subjects who are unlikely to comply with the protocol (eg, have an uncooperative attitude, an inability to return for follow-up visits, or are unlikely to complete the study)
* Subjects who have known impaired hepatic function
* Subjects who have known impaired renal function

AECB-Specific Exclusion Criteria:

* Subjects with acute bronchitis
* Subjects with a known diagnosis of bronchiectasis; cystic fibrosis; lung cancer or lung metastases; or active pulmonary tuberculosis.

CAP-Specific Exclusion Criteria:

* Subjects with severe pneumonia (as defined by the investigator's clinical judgment)
* Subjects with CAP symptoms that require parenteral antibiotic treatment, such as 1 or more of the following conditions:

  * Respiratory frequency >30 breaths/minute
  * Chest x-ray showing an increase in the size of the opacity by ≥ 50% within 48 hours of the initial or current evaluation
  * Shock (systolic blood pressure < 90 mmHg or diastolic blood pressure < 60 mmHg)
  * Altered mental status (disorientation to person, place, or time that is not known to be chronic, lethargy, stupor, or coma)
  * < 90% O2 saturation (by pulse oximetry), or a PaO2 < 60 mmHg
  * Requires mechanical ventilation
  * Requires vasopressors for > 4 hours
  * Urine output < 20 mL/hr or total urine output < 80 mL in 4 hours, unless another explanation is available, or acute renal failure requiring dialysis
  * Hypothermia, defined as core body temperature of < 35°C (95°F)

The investigator and sponsor must approve any waiver of these inclusion and exclusion criteria on a case-by-case basis prior to enrolling a subject. Both the investigator and sponsor must document any waivers.

No subject will be allowed to enroll in this study more than once.

Subjects of Reproductive Potential:

Women of childbearing potential may participate in the study only if the following conditions are met:

* Had a normal menstrual flow ≤ 1 month before study entry
* Has a negative pregnancy test (serum β-subunit hCG) immediately before study entry (ie, before the start of treatment or any other study procedure that could potentially harm the fetus). If obtaining the serum pregnancy test result will cause a delay in treatment, a subject may be entered on the basis of a negative urine pregnancy test sensitive to at least 50 mU/mL, pending results of the serum pregnancy test. Subsequently, if the result of the serum test is positive, the subject must be discontinued from study drug, and every attempt must be made to follow such subjects to term.
* Must agree to use an accepted method of contraception (ie, oral or implanted contraceptive with a barrier method; spermicide and barrier methods; or intrauterine device). The subject must agree to continue with the same method throughout the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2051 (Actual)
Dates: Start 2004-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Post-treatment utilization of healthcare resources, as assessed by unscheduled nonprotocol return office visits, emergency room (ER) visits, hospitalization, and additional nonprotocol antibiotic prescriptions in the 30 days following treatment. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, BS, MT (ASCP), Study Director — Sanofi
Locations (2):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Québec, Canada